CLINICAL TRIAL: NCT06371664
Title: Does the Use of a 3-mm Extended Tray During an At-home Bleaching Treatment Increases Gingival Irritation Associated With This Procedure in an Adult Patient: Randomized Clinical Trial
Brief Title: Gingival Irritation Due to Bleaching Tray Design in an At-home Bleaching Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Patricia Pereira-Lores, Principal Investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023/02
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Gingival Inflammation
Keywords: Tooth bleaching; Vital Bleaching; At-Home bleaching; Gingival Irritation; Bleaching tray
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind clinical trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conventional Tray (1 mm) (Placebo Comparator): Patients put in their individualized 1 mm bleaching trays the bleaching treatment every day during three weeks.
  Interventions: Drug: Conventional Tray (1 mm)
- Extended Tray (3 mm) (Experimental): Patients put in their individualized 3 mm bleaching trays the bleaching treatment every day during three weeks.
  Interventions: Drug: Extended Tray (3 mm)

INTERVENTIONS:
Drug: Conventional Tray (1 mm) — General examination with bite-wings. Dental prophylaxis (dental scaling and polishing with an abrasive paste). Alginate impressions of both arches. Creation of conventional individualized bleaching trays (trimmed 1 mm above the gingival margin) and a position-finder tray of both arches. Application of the bleaching gel in the bleaching trays during 6-8 hours
  Arms: Conventional Tray (1 mm)
Drug: Extended Tray (3 mm) — General examination with bite-wings. Dental prophylaxis (dental scaling and polishing with an abrasive paste). Alginate impressions of both arches. Creation of extended individualized bleaching trays (trimmed 3 mm above the gingival margin) and a position-finder tray of both arches. Application of the bleaching gel in the bleaching trays during 6-8 hours
  Arms: Extended Tray (3 mm)

SUMMARY:
The primary aim of this study is to assess whether the design of the bleaching tray used in at-home bleaching treatment is directly correlated with the risk of gingival irritation. Additionally, it aims to investigate whether the design influences the likelihood of dental sensitivity and its impact on the degree of tooth whitening.

DETAILED DESCRIPTION:
Visit 1: Study information and delivery of informed consent. Recording of the patient's medical history, general examination, and prophylaxis. Alginate impressions will be taken of the upper and lower arches for all patients who meet the inclusion criteria. The impressions will be poured into plaster, and individualized bleaching trays will be made for each patient according to the predetermined assignment ( 1mm extended or 3 mm extended bleaching tray). A positioning guide tray will be fabricated for color measurement.

Visit 2: Initial color measurement with a spectrophotometer and the positioning guide. Each patient will receive their individualized trays. Additionally, they will be given 3 syringes of bleaching agent (Opalescence 16%, Ultradent Products). Each patient will be provided with an instruction sheet and recording sheets to fill out daily during the 3-week study period. They will record if they had gingival irritation and the degree of dental sensitivity.

Visit 3: First-week bleaching review. Data collection (gingival irritation + color + sensitivity).

Visit 4: Second-week bleaching review. Data collection (gingival irritation + color + sensitivity).

Visit 5: Third-week bleaching review and end of the study. Data collection (gingival irritation + color + sensitivity).

ELIGIBILITY:
Inclusion Criteria:

* No oral or systemic pathology
* Periodontally healthy
* No cavities
* Tooth shade of the upper and lower canines A2 or darker

Exclusion Criteria:

* Adhesive restorations or prostheses in the anterior region
* Enamel or dentin alterations
* Smoking
* Pregnant women
* Undergone prior bleaching treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Subjective questionnaire of gingival irritation | Daily, during 3 weeks
  Patients should answer daily a dental sensitivity questionnaire. They should mark a "0" if their gingival tissue appeared normal or a "1" If they observed GI, defined as the presence of a white or red layer on the gingiva.Patients who scored "0" during the treatment were classified as individuals without gingival irritation.
Objective clinical examination of gingival irritation | Once a week, during 3 weeks
  Clinicians examined visually and with a periodontal probe the gingival tissue.Patients were categorized according to Löe and Silness' gingival index as: G0 (normal gingiva); G1(mild inflammation: slight change in color, slight edema; no bleeding on probing); G2 (moderate inflammation: redness, edema and glazing; bleeding on probing); and G3 (severe inflammation: marked redness and edema; ulceration; tendency to spontaneous bleeding).Patients will a score of 0 during the treatment will be defined as patients with no gingival irritation. The individual highest recorded score will be the grade of gingival irritation.

SECONDARY OUTCOMES:
Questionnaire of dental sensitivity | Daily, during 3 weeks
  Patients should answer a dental sensitivity questionnaire. A a 5-point subjective numerical classification scale will be used (0=no sensitivity, 1=light, 2=mild, 3=considerable and 4=severe). Patients will a score of 0 during the treatment will be defined as patients with no sensitivity. The individual highest recorded score will be the grade of intensity for each patient.
Shade evaluation with a dental spectrophotometer | Once a week, during 3 weeks
  The color will be measured with a dental spectrophotometer and the parameters L (Lightness), C (Chroma) and H (Hue) will be recorded. To determine the color change between visits the CIEDE2000 formula will be used.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Medicine and Dentistry, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pereira-Lores P, Martin-Gonzalez J, Gancedo-Gancedo T, Alonso de la Pena V, Alvarez-Novoa P, Varela-Aneiros I, Abella-Sans F, Martin-Biedma B, Castelo-Baz P. Does the use of a 3-mm extended tray during an at-home bleaching treatment increase gingival irritation? A randomized clinical trial. J Prosthet Dent. 2025 May;133(5):1277-1283. doi: 10.1016/j.prosdent.2024.09.029. Epub 2024 Nov 18. PMID 39562219